CLINICAL TRIAL: NCT06794788
Title: Effect of Immersive Virtual Reality on Pain in Different Dental Procedures in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Research Grant No: 20190440; Research Grant No: 20190440 (Other Grant/Funding Number: Jordan University of Science and Technology)
Record Dates: First submitted 2025-01-16; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Fissure Sealant; Space Maintainer; Impression Taking for Space Maintainers; FLUORIDE THERAPY; SCALING; Stainless-steel Crown; Pulp Therapy; Restorations; TOOTH Extraction
Keywords: VIRTUAL REALITY; PAIN; DENTAL
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GROUP A1 (No Intervention): The children with dental procedures not requiring administration of LA were assigned to Group A. Divide the children in Group A into two sub-groups(Group A1 & A2) Patients included in Group A1 randomly assigned to receive no VR
- GROUP A2 (Experimental): The children with dental procedures not requiring administration of LA were assigned to Group A. Divide the children in Group A into two sub-groups(Group A1 & A2) Patients included in Group A2 randomly assigned to receive VR-The iWear
  Interventions: Device: VR-The iWear
- GROUP B1 (No Intervention): the children with dental procedures requiring administration of LA were assigned to Group Divided the children in Group B into two sub-groups (Group B1 & B2) Patients included in Group B1 randomly assigned to receive no VR
- GROUP B2 (Experimental): the children with dental procedures requiring administration of LA were assigned to Group Divided the children in Group B into two sub-groups (Group B1 & B2) Patients included in Group B2 randomly assigned to receive VR-The iWear
  Interventions: Device: VR-The iWear

INTERVENTIONS:
Device: VR-The iWear — The immersive virtual reality device was used for this study from(Vuzix®, Rochester, New York, USA). The iWear consists of a lightweight high-end pair of video headphones that contain pair of VR goggles
  Arms: GROUP A2; GROUP B2

SUMMARY:
the current study aims to assess virtual reality as an effective pain management technique for children undergoing different dental procedures.

The iWear is the immersive virtual reality device was used for this study from (Vuzix®, Rochester, New York, USA). The iWear consists of a lightweight high-end pair of video headphones that contain pair of VR goggles

DETAILED DESCRIPTION:
The peadiatric dentist examined children to assess their needs. At the screening, a full mouth oral examination was performed. Different dental procedures needed were determined based on the outcome of the clinical examination performed. Some of these dental procedures did not require administration of local anesthesia (LA), such as fissure sealant, space maintainer, fluoride therapy, impression taking for space maintainers, and scaling. Other dental procedures require the administration of LA , such as stainless-steel crown, pulp therapy, restorations, and extraction (Figure 2). The peadiatric dentist divided the children into two groups (Group A & B) according to the need for usage of LA. The children with dental procedures not requiring administration of LA were assigned to Group A, and the children with dental procedures requiring administration of LA were assigned to Group B. A computer-generated random number was used to randomly divide the children in Group A into two sub-groups(Group A1 & A2) according to the usage of VR. Patients included in Group A1 randomly assigned to receive no VR. On the other hand, patients included in Group A2 randomly assigned to receive VR. Also, children in Group B were randomly assigned into two sub-groups (Group B1 & B2) to receive no VR or VR respectively.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 5-12 years
* Good general health,
* Taking no medications,
* Willingness to participate in the study

Exclusion Criteria:

* Subjects with a convulsive disorder,
* Subjects with a history of serious vestibular abnormalities,
* Subjects with musculoskeletal disorders, or developmental delay taking psychotropic drugs

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
The Wong-Baker Faces | through study completion, an average of 2 years
  used to measure the level of pain in the current study. The Wong-Baker Faces is a self-report measure that consists of six cartoon faces with different facial expressions. The Wong-Baker Faces scale starts from zero to 10
Visual Analog Scale (VAS) | through study completion, an average of 2 years
  The VAS is a self-report measure that consists of a 10-centimeters horizontal line that indicates the current level of pain. The children were asked to give ratings using 0-10 scales with lower numbers indicates less pain, while the higher numbers indicate higher pain.
The 'Face, Legs, Activity, Cry, Consolability' (FLACC) scale | through study completion, an average of 2 years
  s a behavioral pain observation scale used commonly to measure pain during a procedure. The FLACC are reliable and valid common pain measurement tool used as an external evaluator to measure procedural pain.
  Each category is scored on a 0-2 scale, resulting in a total 0-10 score. The external evaluator used a 0-10 scale, with cut points indicating (0) Relaxed, (1-3) Mild discomfort, (4-6) Moderate pain, or (7-10) Severe discomfort/pain

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: JANUARY 2025 TILL MAY 2025
Access Criteria: ANYONE ASKING FOR THE INFROMATION.IT WILL BE PROVIDED THROUGH A LINK AND IT WILL BE RAW DATA
URL: https://doi.org/10.6084/m9.figshare.27124410.v1

REFERENCES:
- [Background] Al-Khotani A, Bello LA, Christidis N. Effects of audiovisual distraction on children's behaviour during dental treatment: a randomized controlled clinical trial. Acta Odontol Scand. 2016 Aug;74(6):494-501. doi: 10.1080/00016357.2016.1206211. Epub 2016 Jul 13. PMID 27409593
- [Background] Hoffman HG, Patterson DR, Carrougher GJ. Use of virtual reality for adjunctive treatment of adult burn pain during physical therapy: a controlled study. Clin J Pain. 2000 Sep;16(3):244-50. doi: 10.1097/00002508-200009000-00010. PMID 11014398
- [Background] Felemban OM, Alshamrani RM, Aljeddawi DH, Bagher SM. Effect of virtual reality distraction on pain and anxiety during infiltration anesthesia in pediatric patients: a randomized clinical trial. BMC Oral Health. 2021 Jun 25;21(1):321. doi: 10.1186/s12903-021-01678-x. PMID 34172032
- [Background] Koticha P, Katge F, Shetty S, Patil DP. Effectiveness of Virtual Reality Eyeglasses as a Distraction Aid to Reduce Anxiety among 6-10-year-old Children Undergoing Dental Extraction Procedure. Int J Clin Pediatr Dent. 2019 Jul-Aug;12(4):297-302. doi: 10.5005/jp-journals-10005-1640. PMID 31866714
- [Background] Klingberg G, Broberg AG. Dental fear/anxiety and dental behaviour management problems in children and adolescents: a review of prevalence and concomitant psychological factors. Int J Paediatr Dent. 2007 Nov;17(6):391-406. doi: 10.1111/j.1365-263X.2007.00872.x. PMID 17935593
- [Background] Grisolia BM, Dos Santos APP, Dhyppolito IM, Buchanan H, Hill K, Oliveira BH. Prevalence of dental anxiety in children and adolescents globally: A systematic review with meta-analyses. Int J Paediatr Dent. 2021 Mar;31(2):168-183. doi: 10.1111/ipd.12712. Epub 2020 Sep 9. PMID 33245591